CLINICAL TRIAL: NCT04424719
Title: Follow-up of Patients With Uveal Melanoma Adapted to the Risk of Relapse (SALOME)
Acronym: SALOME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IC2019-13
Record Dates: First submitted 2020-05-18; First posted 2020-06-11 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-07

CONDITIONS: Uveal Melanoma
Keywords: uveal melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Hematologic Tests; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with uveal melanoma (Other): High risk patients are referred for the medical oncology consultation to organize oncological surveillance after general staging of the disease. For enucleated patients, a blood sample is required according to the study schedule.
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — High risk patients are referred for the medical oncology consultation to organize oncological surveillance after general staging of the disease. Signature of the informed consent of SALOME study, inclusion in the study and risk-adjusted surveillance schedule :
  (i) Liver MRI every 6 months performed at the expert center for UM (according to guidelines).
  (ii) For enucleated patients, a blood sample (3 x 6 ml EDTA tubes) is taken every 6 months according to the schedule below. Plasma and mononucleated cells will be isolated and preserved for bio-markers research.
  * M0 : during the first medical oncology visit.
  * At each imaging assessment, every 6 months for at least 5 years (M6 to M60) and 10 years maximum (M120).
  * At the diagnosis of metastasis.
  * At each significant event during the metastatic disease (surgery, treatment response or progression).
  Other Names: MRI in routine

SUMMARY:
Biomarkers search for early diagnosis of liver metastases in patients with uveal melanoma who benefit from a follow-up tailored to their personalized risk of relapse.

DETAILED DESCRIPTION:
High risk patients are referred for the medical oncology consultation to organize oncological surveillance after general staging of the disease. Signature of the informed consent of SALOME study, inclusion in the study and risk-adjusted surveillance schedule :

(i) Liver MRI every 6 months performed at the expert center for UM (according to guidelines).

(ii) For enucleated patients, a blood sample (3 x 6 ml EDTA tubes) is taken every 6 months according to the schedule below. Plasma and mononucleated cells will be isolated and preserved for bio-markers research.

* M0 : during the first medical oncology visit.
* At each imaging assessment, every 6 months for at least 5 years (M6 to M60) and 10 years maximum (M120).
* At the diagnosis of metastasis.
* At each significant event during the metastatic disease (surgery, treatment response or progression).

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged of 18 years or more.
2. Patient with uveal melanoma with high metastatic relapse risk defined as :

   * T2b/c/d ou ≥ T3,
   * or chromosom 3 or chromosom 8 abnormality by CGH array.
3. Completion of treatment of the primary tumor ≤ 2 months.
4. Patient able to comply with the schedule of visits and blood samples of the study.
5. Signed informed consent form or legal representative.

Exclusion Criteria:

1. Patient without french social insurance.
2. Any social, medical or psychological condition making the research process impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2037-07-07 (Estimated); Study Completion 2037-07-07 (Estimated)

PRIMARY OUTCOMES:
Description of the metastatic events and treatments in high risk UM patients and correlation to biomarkers | 120 months
  metastatic events and treatments reports correlation with their ocrresponding biomarquers
Biological study (lymphocytes) | 120 months
  lymphocyte phenotype analysis with biological tests
Biological study (ctDNA) | 120 months
  circulating tumor DNA analysis with biological tests

SECONDARY OUTCOMES:
Biological samples prospective collection (ctDNA) | 120 months
  collection of biological samples (circulating tumor DNA analyses)
Biological samples prospective collection (immune-monitoring analyses) | 120 months
  collection of biological samples (immune-monitoring analyses) with biological tests
Biological samples prospective collection (sequencing analyses) | 120 months
  collection of biological samples (sequencing analyses) with biological tests
Comparison of clinical and imaging data (MRI) | 120 months
  Comparison of imaging data (MRI) between the patients with and without identified biomarkers (biological tests)
Comparison of clinical and imaging data (clinical data) | 120 months
  Comparison of clinical data between the patients with and without identified biomarkers (biological tests)
Univariate analysis of the prognostic value of identified biomarkers | 120 months
  prognostic value of identified biomarkers analysis with biological tests
Multivariate analysis of the prognostic value of identifies biomarkers adjusted for clinical and imaging data | 120 months
  Multivariate analysis of the prognostic value of identifies biomarkers (biological tests) adjusted for clinical (medical patients records) and imaging data (MRI)
Analysis of discordant cases regarding genomic/tumor size prognostic factors and outcomes | 120 months
  Analysis of discordant cases regarding genomic/tumor size prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Piperno-Neumann, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).